CLINICAL TRIAL: NCT02706860
Title: Efficacy of Different Perioperative Statin Regimens on the Protection Against Post Coronary Artery Bypass Grafting Major Adverse Cardio-cerebral Events
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Elmarsafawi, Teaching Assistant, Clinical Pharmacy Department, Faculty of Pharmacy, Cairo University), Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CL (775)
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Bypass Grafting
MeSH Terms: interventions — Atorvastatin

ARMS (3):
- "80 mg atorvastatin for 2 days" regimen (Experimental): 80 mg atorvastatin/ day for 2 days before coronary artery bypass grafting. This dose was restarted postoperative and continued for 1 month.
  Interventions: Drug: Atorvastatin
- "40 mg atorvastatin for 5-9 days preoperative" regime (Experimental): 40 mg atorvastatin/ day for 5-9 days before coronary artery bypass grafting. This dose was restarted postoperative and continued for 1 month.
  Interventions: Drug: Atorvastatin
- "80 mg atorvastatin for 5-9 days preoperative" regime (Experimental): 80 mg atorvastatin/ day for 5-9 days before coronary artery bypass grafting. This dose was restarted postoperative and continued for 1 month.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
This study aims at comparing different perioperative statin regimens for the prevention of post CABG adverse events.

This was a randomized, prospective clinical trial. Ninety four patients scheduled for elective, isolated on- or off- pump CABG were randomly assigned to one of 3 treatment groups; 80 mg atorvastatin/day for 2 days preoperatively (N=37), 80 mg atorvastatin/day for 5-9 days preoperatively (N=28) or 40 mg atorvastatin/day for 5-9 days preoperatively (N=29). The corresponding preoperative doses were restarted postoperatively (post-op) when patients were able to take the medication orally and were continued for one month. Cardiac troponin I (TnI), Creatine Kinase (CK-MB) and C-reactive protein (CRP) were assayed preoperatively and post-operatively at 8, 24, 48 hours, and at discharge. Marker levels were compared among the three groups. The incidence of post-operative major adverse cardiac and cerebrovascular events (MACCE) was assessed including; 30-day all-cause mortality, myocardial infarction, atrial fibrillation, ventricular tachycardia/ventricular fibrillation, stroke and target-vessel revascularization. The incidence of renal or hepatic impairment and post-operative infections were also assessed. A Quality of life (QoL) questionnaire (EQ-5D-3L) was administered preoperatively and 1 month after CABG.

DETAILED DESCRIPTION:
This study was conducted at the National Heart Institute (NHI), Cairo, Egypt, during the period between June 2013 and February 2015. It was approved by the ethics committee at the Faculty of Pharmacy, Cairo University, and the scientific committee at the NHI. An informed consent was obtained from all study participants after they have been approached with the nature, purpose and possible risks of the study.

Preoperative baseline demographic characteristics, preoperative medications, comorbid conditions and risk factors were identified and summarized.

Design: This is a randomized, prospective, interventional, open label study. Upon admission to the NHI, eligible patients were randomly assigned to one of 3 treatment groups; group I (80 mg atorvastatin/day for 2 days preoperatively), group II (40 mg atorvastatin/day for 5-9 days preoperatively) or group III (80 mg atorvastatin/day for 5-9 days preoperatively). Atorvastatin doses were reinitiated postoperatively as soon as patients could take the medication orally and was continued for one month after operation.

The following intra-operative data were recorded for each patient; cardiopulmonary bypass time, aortic clamp time, type of anesthesia, number of grafts and need for blood transfusion.

Blood samples were drawn preoperatively (baseline) then at 8 hours, 24 hours, 48 hours postoperatively and before hospital discharge. Blood samples were spun and sera were separated, stored according to the storage conditions specified by the manufacturer, and used to measure the TnI, CK-MB and CRP at the time of analysis. Cardiac TnI was assayed by the Dimension® TNI method, a homogenous sandwich chemiluminescent assay based on LOCI® technology, using SIEMENS Dimension® EXL™, LOCI® Module system. Siemens Healthcare Diagnostics Inc. Newark, USA. CK-MB isoenzyme was measured by the Mass MMB method, a one-step enzyme immunoassay based on the sandwich principle, using SIEMENS Dimension® Heterogeneous Immunoassay Module system. Siemens Healthcare Diagnostics Inc. Newark, USA. CRP was measured by the C-Reactive Protein Extended Range (RCRP) method, a method based on a particle enhanced turbidimetric immunoassay (PETIA) technique, using SIEMENS Dimension® system. Siemens Healthcare Diagnostics Inc. Newark, USA.

A-12 lead electrocardiogram (ECG) was performed pre-operatively, in the intensive care unit (ICU) and upon patient transfer to the ward. The appearance of new Q-waves indicating myocardial infarction (MI) or incidence of any arrhythmias was reported. Echocardiography was performed pre-operatively and post-operatively after ICU discharge to detect any new wall movement abnormalities as well.

Measured end points were as follows: 1) Incidence of post-operative major adverse cardiac and cerebrovascular events (MACCE) including; 30-days all-cause mortality, MI, AF, ventricular tachycardia or ventricular fibrillation, debilitating stroke or transient ischemic attack (TIA) or target-vessel revascularization; 2) renal impairment; 3) hepatic impairment; 4) postoperative infections; 5) persistent blood glucose abnormalities; 6) length of ICU and hospital stays, and a health-related quality-of-life (HRQoL). HRQoL was assessed using the Euro Quality of Life 5-Dimensional Classification (EQ-5D-3L) 19 at baseline (preoperatively) as patients were admitted to the NHI and then one month postoperatively during the follow-up visit or by contacting the patient via a phone call.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic Heart Disease patients referred for elective isolated on- or off- pump CABG
* Adult patients with normal preoperative hemoglobin, hematocrit, albumin, cardiac markers; Cardiac troponin I (TnI) and Creatine Kinase-MB (CK-MB) levels.
* Serum creatinine < 2 mg/dl and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times upper normal limit (UNL).

Exclusion Criteria:

* Recent history of stroke, myocardial infarction (MI), atrial fibrillation (AF) or any other type of arrhythmias.
* Any malignancy, inflammatory or muscle disease were not included in this study.
* Hypersensitivity to statins or on medications that are known to interact with statins.

Ages: 42 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative major adverse cardiocerebral events | 30 days